CLINICAL TRIAL: NCT00188422
Title: Surveillance Low Dose Computed Tomography of the Thorax in Patients With High Grade Extremity Soft Tissue Sarcoma
Brief Title: Study of Low Dose CT in Sarcoma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 03-0468-CE
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2007-04-23 (Estimated); Status verified 2007-04

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma

INTERVENTIONS:
Procedure: low dose CT

SUMMARY:
The primary outcome of this study is the detection of lung metastases comparing Low dose CT (LDCT) and Minimum dose CT (MnDCT) with CXR.

Hypothesis

1. LDCT and MnDCT have similar sensitivity for the detection of lung nodules (metastases).
2. MnDCT of the thorax detects a larger number of nodules (metastases) than CXR.

DETAILED DESCRIPTION:
A 3-year prospective phase II non-randomized study commenced May 2003 enrolling 60 high-risk patients with Intermediate and High Grade STS. Each patient is kept under radiological surveillance for 3 years unless lung metastases are detected. Conventional thoracic imaging for staging and surveillance of STS patients is shown in Figure 1. In the trial, LDCT and MnDCT are added to each imaging visit (Figure 1). A 2-view CXR (CR) is performed (Direct View, Kodak, Rochester) followed by thoracic CT scans performed on a Siemens 16 row MDCT (Sensation 16, Siemens, Erlangen), CT acquisition; 120kVp, 5/2.5/2.5mm. Images are reconstructed with high and low spatial frequency filters and soft copy viewing is performed on a standalone PACS workstation using standard mediastinal (w 350, l 40) and lung (w 1500, l -600) settings. Examinations are performed with varying mAs; SDCT 120 mAs, LDCT 40 mAs and MnDCT 20 mAs. The examinations are evaluated, blinded to the results of the alternative and previous studies, for the presence of nodules (defined as a non-calcified focal opacity ≥3 mm < 3 cm). Surveillance imaging is commenced 3 months post surgery.

ELIGIBILITY:
Inclusion Criteria:

* High Grade Soft tissue sarcoma

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70
Dates: Start 2003-08; Study Completion 2006-01

PRIMARY OUTCOMES:
Detection of metastases

CONTACTS AND LOCATIONS:
Overall Officials: Narinder Paul, FCPC C, Principal Investigator — University Health Network, Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada